CLINICAL TRIAL: NCT01219010
Title: A Study of Siltuximab (Anti-IL-6 Monoclonal Antibody) Effects on the QT Interval in Subjects With Monoclonal Gammopathy of Undetermined Significance, Smoldering Multiple Myeloma, or Indolent Multiple Myeloma
Brief Title: A Study Evaluating the Effects of Siltuximab on the Heart in Patients With Monoclonal Gammopathy of Undetermined Significance, Smoldering Multiple Myeloma, or Indolent Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017452; CNTO328SMM1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-09-23; First posted 2010-10-13 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma; Plasma Cell Neoplasm
Keywords: Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma; Indolent Multiple Myeloma; QT; Siltuximab; CNTO 328; IL-6; Monoclonal Antibody
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma; Neoplasms, Plasma Cell; Smoldering Multiple Myeloma | interventions — siltuximab

ARMS (1):
- 001 (Experimental): Siltuximab 15mg/kg IV infusion every 3 weeks for 4 cycles. If applicable extended dosing of 15 mg/kg IV infusion every 4 weeks for up to 2 years.
  Interventions: Biological: Siltuximab

INTERVENTIONS:
Biological: Siltuximab — 15mg/kg IV infusion every 3 weeks for 4 cycles. If applicable extended dosing of 15 mg/kg IV infusion every 4 weeks for up to 2 years.

SUMMARY:
The purpose of this study is to determine if siltuximab has an effect on the heart function measured by ECG recordings and more specifically to determine if siltuximab has an effect on the QT interval in patients with Monoclonal Gammopathy of Undetermined Significance (MGUS), Smoldering Multiple Myeloma (SMM) or Indolent Multiple Myeloma (IMM). The study will also look to see if siltuximab may be useful in treating patients with MGUS, SMM or IMM.

DETAILED DESCRIPTION:
This is a research study with an experimental drug called siltuximab (also known as CNTO 328). Currently there are studies with siltuximab, completed or ongoing, in patients with blood cancers such as multiple myeloma and Castleman's disease and with solid tumors such as kidney, ovarian and prostate cancer, to see if siltuximab is safe and to determine what effects it has on these types of cancer. This study is being done in patients with Monoclonal Gammopathy of Undetermined Significance (MGUS), Smoldering Multiple Myeloma (SMM) or Indolent Multiple Myeloma (IMM) to determine if siltuximab has an effect on heart function measured by ECG recordings, and more specifically to determine if siltuximab has any effect on the QT interval. MGUS, SMM and IMM patients usually go on to develop active multiple myeloma which is a type of cancer that affects the blood and bone marrow. The cancer cells in the bone marrow can cause the normal bone marrow cells to breakdown. This can result in low levels of red blood cells (which may make the patient feel tired or fatigued), low levels of white blood cells (which may increase the patient's chances of infections) or low levels of platelets (which may increase risk of bleeding). The cancer cells can cause damage to the normal bone. This can cause bone pain, bone fractures, and can increase the level of calcium in the blood. The cancer cells also make proteins (called M-proteins), which can result in damage to other organs, especially the kidneys. Siltuximab is a chimeric (part mouse and part human) antibody (immunoglobulin that is important for fighting infection). It does this by blocking another small protein called Interleukin 6 (IL-6). The body makes IL-6 naturally, and at normal levels it is important for the inflammatory response. But high levels of IL-6 can help cancer cells grow and interfere with chemotherapy drugs killing cancer cells. Cancer-related sicknesses such as weight loss, bone weakening, and depression have been linked to high levels of IL-6. This study will also look to see if siltuximab may be useful in treating patients with MGUS, SMM or IMM. All participating patients will be in the study for about 6 months and will receive siltuximab four (4) times every 3 weeks at a dose of 15mg per kg bodyweight. Siltuximab is given as a 1 hour intravenous infusion, through a small tube that goes directly into the vein. Following this treatment period, patients showing a response, defined as a 50% or higher reduction in M-protein in their blood/urine, may be allowed to continue treatment with siltuximab 15mg/kg every 4 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MGUS (measurable serum M-protein < 3 g/dL AND clonal bone marrow plasma cells < 10% without any end organ damage), SMM (measurable serum M-protein = 3 g/dL OR clonal bone marrow plasma cells = 10% without any end organ damage) or IMM (measurable serum M-protein = 3 g/dL OR clonal bone marrow plasma cells = 10% and = 3 lytic bone lesions but no other end organ damage)
* Qualifying ECG results that will be checked by a central laboratory
* Negative urine drug screen for substances of abuse
* Qualifying hematology and chemistry laboratory results.

Exclusion Criteria:

* Diagnosis of symptomatic multiple myeloma
* Prior exposure to approved or investigational myeloma treatments
* Prior exposure to agents targeting IL-6 or the IL-6 receptor
* Significant cardiac disease
* Skin condition likely to interfere with ECG electrode placement, breast implant, or thoracic surgery
* Received medications known to affect the QT interval
* Vaccination with live, attenuated vaccines within 4 weeks
* Major surgery or radiation within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
QTc interval | Screening through Week 10

SECONDARY OUTCOMES:
Additional safety evaluations | 6 months and, if eligible, up to 2 years of extended treatment
Efficacy evaluations | 6 months and, if eligible, up to 2 years of extended treatment
Pharmacokinetic and Pharmacodynamic evaluations | 6 months and, if eligible, up to 2 years of extended treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- United States (3):
  - Chicago, Illinois
  - Dallas, Texas
  - Houston, Texas
- Belgium (2):
  - Antwerp
  - Ghent
- Russia (3):
  - Izhevsk
  - Moscow
  - Nizhny Novgorod

REFERENCES:
- See also: A Study of Siltuximab (Anti-IL-6 Monoclonal Antibody) Effects on the QT Interval in Subjects with Monoclonal Gammopathy of Undetermined Significance, Smoldering Multiple Myeloma, or Indolent Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=213&filename=CR017452_CSR.pdf